CLINICAL TRIAL: NCT04228575
Title: Optimizing Duration of Therapist-guided Internet-delivered Cognitive Behaviour Therapy for Anxiety and Depression
Brief Title: Optimizing Duration of Therapist-guided Internet-delivered Cognitive Behaviour Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2019-197
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; internet-delivered cognitive behaviour therapy; randomized controlled trial; patient-centred; personalized therapy; knowledge implementation; mental health system; therapist-assistance; booster session; factorial design
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Extended Contact (Experimental): Clients in the Extended Contact condition will be asked at the 6 week mark if they like they can extend their treatment and receive up to 12 weeks of support. They will be informed that this may be helpful if they feel they have fallen behind in reviewing of the materials, if they would like to receive support while they work on supplementary resources or if they would like extended support while they work on core lessons. If they would like additional support, participants will answer questions presented on the website about their desire for this additional support what they would like to focus on during this time. Those clients who indicate that they would like this extended support will automatically have their therapists check-in with them for up to 12 weeks. Those that do not request the additional support will end treatment as planned at the end of 8 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- 8 Week ICBT no Booster (Experimental): In the standard condition, clients will receive 8 weeks of therapist support. They will not be given the option to extend their treatment and support to 12 weeks. The booster course will not be offered in this condition.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- Extended Contact with Booster (Experimental): Clients in the Extended Contact condition will receive an email at the 6 week mark letting them know that they if they like they can extend their treatment and receive up to 12 weeks of support. At week 6, clients will answer questions on the website about whether they would like this additional support or not and what they would like to focus on during this time. Clients who indicate they would like this extended support will automatically have their therapists check-in with them for up to 12 weeks.
  They will also be told that at 16 weeks they will have access to a booster session (online materials that go over core skills such as thought challenging, deep breathing, behavioural activation, and graded exposure). At 16 weeks, they will be sent an email reminder to log in for the booster course. The therapist will send a supportive email to the client offering to assist with any challenges the client reports in the check-in questionnaire by email or phone call over the next 2 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy
- 8 week ICBT with Booster (Experimental): Clients in the booster condition will be told that at 16 weeks they will have access to a booster session (online materials that go over core skills such as thought challenging, deep breathing, behavioural activation, and graded exposure). At 16 weeks, they will be sent an email reminder to log in for the booster course. The therapist will send a supportive email to the client offering to assist with any challenges the client reports in the check-in questionnaire by email or phone call over the next 2 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behaviour therapy

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behaviour therapy — All clients will receive the Wellbeing Course developed at Macquarie University, Australia. The Wellbeing Course is a transdiagnostic Internet-delivered cognitive behaviour intervention targeting symptoms of depressive and anxiety disorders. It comprises 5 online lessons targeting: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure; and 5) relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills) and include homework activities. Lessons are released gradually in a standardized order over 8 weeks. Phone calls will only be made if there is a significant clinical issue requiring therapist attention that cannot be addressed over email (e.g., sudden increase in symptoms). Therapists will spend ~15 mins. per week/per client.

SUMMARY:
Depression and anxiety are common and prevalent conditions that are frequently under treated. In an attempt to increase timely and accessible psychological treatment, Internet-delivered Cognitive Behaviour Therapy (ICBT) has emerged. ICBT involves delivering therapeutic content to manage depression and or anxiety via structured online lessons. This is often combined with brief therapist guidance, for example once per week for 8 weeks via secure messaging or phone calls. Although outcomes of ICBT are very impressive, there is room for improvement in terms of completion rates and outcomes. Feedback from patients suggest that some patients would prefer longer term support or follow-up care.

In this two-factorial randomized controlled trial, the investigators aim to contribute to the literature by examining whether the efficacy of ICBT is improved by offering an extended period of support to clients (from 8 weeks to 12 weeks) and being offered a booster session at 16 weeks after treatment enrollment (yes vs no). Follow-up assessments will be conducted at 8, 16 and 26 weeks after treatment enrollment. Primary outcomes are reduced anxiety and depression. Secondary outcomes include reduced panic, social anxiety, trauma, quality of life, disability, work productivity, and healthcare use.

DETAILED DESCRIPTION:
Past research of ICBT offered in routine care has found that patients and therapists often recommend "personalizing" the delivery of ICBT, for example, by increasing the length of time therapist support is available or offering booster sessions after treatment has ended. To date, in terms of ICBT, there has been limited research on the impact of extending support after treatment materials have been delivered or offering a booster session.

In this trial, the investigators will examine if the efficacy of ICBT is improved by offering an extended period of support to clients (from 8 weeks to 12 weeks) or by being offered a booster session at 16 weeks after treatment enrollment (yes vs no). Follow-up assessments will be conducted at 8, 16 and 26 weeks after treatment enrollment. Primary outcomes are reduced anxiety and depression. Secondary outcomes include reduced panic, social anxiety, trauma, quality of life, disability, work productivity, and healthcare use. The impact of these factors on intervention usage (e.g., completion rates, log-ins, emails sent) and treatment satisfaction will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Endorse symptoms of anxiety or depression
* Resident of Saskatchewan
* Access to a computer and the Internet

Exclusion Criteria:

* Have a severe psychiatric illness (e.g. psychosis)
* Assessed as being at high risk of suicide
* Report severe problems with alcohol or drugs
* Report severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline (Screening), weeks 1-12, 16 and 26 week from enrollment
  Change in depression symptoms. 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (Screening), weeks 1-12 and 16 and 26 week from enrollment
  Change in anxiety symptoms. 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Panic Disorder Severity Scale Self-report | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Change in panic symptoms. Items are summed into a total score. Total scores range between 0 and 28, with higher scores representing more severe self-reported symptoms of panic.
Social Interaction Anxiety Scale (6 items) | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Change in social anxiety symptoms. Items from the two measures are summed into a total score. Total scores range between 0 and 24, with higher scores representing more severe self-reported symptoms of social phobia
Social Phobia Scale-Short form (6 items) | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Change in social anxiety symptoms. Items from the two measures are summed into a total score. Total scores range between 0 and 24, with higher scores representing more severe self-reported symptoms of social phobia
Quality of Life (EQ-ED-5L) | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Change in quality of life. Items are summed into six sub-total scores. The first five sub-total scores respectively assess various domains of quality of life (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
  Each of the five sub-total scores range between 1 and 5, with higher scores representing greater self-reported severity and impairment in these various domains. The last sub-total score provides an overall index of health and can range between 0 and 100, with higher scores representing better self-reported health.
Mental Health Service Use, Medication, and Employment | Baseline (Screening) and Week 26 week from enrollment
  This measure is 19 items and measures direct and indirect cost of mental health symptoms. Frequency of visits to health specialists (e.g., family doctor, walk-in clinic, psychiatrist, psychologist, social worker, nurse/community nurse/psychiatric nurse) or use of health services (e.g. psychiatric day-patient/part-time treatment, alcohol or drug treatment program, self-help group, ambulance/paramedics, crisis service, hospital admission) in the previous 3 months for mental health reasons are collected. Medication use/changes in previous 3 months for mental health concerns. Questions about occupation, hours in contract, and time off work in previous 3 months for mental health concerns.
Treatment Satisfaction | Week 8, 16 and 26 week from enrollment
  Measure includes 19 questions assessing satisfaction with various aspects of Internet-CBT and also negative effects of treatment
Insomnia Severity Index (ISI) | Baseline
  Measure includes 7 questions rated on a 0-4 point scale with higher scores indicative of higher levels of insomnia.
Sheehan Disability Scale (SDS) | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Higher total scores indicate a greater degree of impairment. Total scores range from 0 to 30. Scores in each of 3 specific life domains range from 0 to 10.
Life Events Checklist for DSM-5 (LEC-5) | Baseline (Screening)
  Life Events Checklist for DSM-5 (LEC-5). A checklist of common traumatic events used to establish the nature of the traumatic events a respondent has experienced. This questionnaire is not intended to be scored but is used for descriptive purposes.
PTSD Checklist for DSM-5 (PCL-5) | Baseline (Screening), week 8, 16 and 26 week from enrollment
  Higher total scores indicate greater severity of posttraumatic stress. Scores range from 0 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada